CLINICAL TRIAL: NCT06506669
Title: Comparing Two Normal Approaches to Procedural Sedation for Cataract Surgery: A Prospective, Feasibility Pilot Study
Brief Title: Cataract Monitored Anesthesia Care (MAC) Feasibility Pilot Study
Acronym: CaTNAPS-1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 23-40367; 5K23AG072035-03 (NIH)
Record Dates: First submitted 2024-06-25; First posted 2024-07-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cataract; Bilateral Senile Cataract; Anesthesia; Patient Satisfaction
Keywords: cataract surgery; oral sedation; intravenous sedation; conscious sedation; monitored anesthesia care; quality of recovery
MeSH Terms: conditions — Cataract; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: A single-center, randomized, double-blinded, randomized pilot clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, clinicians (operating room nurses, ophthalmologists, and anesthesia staff), and research staff responsible for data collection and analysis will be blinded to the treatment group in order to minimize bias and maximize the validity of results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Oral sedation will be administered to patients prior to the procedure.
  Interventions: Procedure: Oral sedation
- Placebo (Placebo Comparator): An oral placebo pill will be administered to patients prior to the procedure.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Oral sedation — Oral medication for anxiolysis administered in the preoperative setting
  Arms: Intervention
Procedure: Placebo — A placebo pill with no active ingredients administered in the preoperative setting
  Arms: Placebo

SUMMARY:
The goal of this pilot clinical trial comparing two different sedation approaches for cataract surgery is to assess patient satisfaction, the quality of recovery, and surgical outcomes as well as to evaluate the overall feasibility and acceptability of the study protocol for the purpose of planning a larger clinical trial. Participants will be asked to respond to several surveys throughout the study on their experience and to assess outcomes of interest.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blinded, pilot clinical trial (n=20). Participants having first eye cataract surgery will be randomized to receive an oral benzodiazepine (intervention) or an oral placebo pill (control). The primary goal of this study is to compare differences in patient satisfaction, quality of recovery and surgical outcomes in participants receiving oral sedation versus oral placebo for cataract surgery. The secondary goals of this study are to assess success with recruitment, intervention fidelity, adherence to interventions and participant retention after interventions. Participants will be asked to respond to several surveys at key study timepoints regarding their sedation experiences and to assess outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 60 years old
2. Capable of providing informed consent and completing the study procedures in English
3. Able to provide consent for oneself
4. Able to follow directions
5. Able to climb one flight of stairs without stopping to rest
6. Have a new diagnosis of cataract disease
7. Plan on having cataract surgery on their eye within the next 6 months

Exclusion Criteria:

1. History of prior cataract surgery
2. Admission to the hospital within the past 30 days
3. Difficulty being sedated during other minor outpatient procedures or imaging studies
4. Allergy or resistance to local anesthetic agents
5. Cannot lay flat on your back without having symptoms (i.e., difficulty breathing, severe back pain, etc.)
6. History of severe anxiety requiring routine use of benzodiazepines
7. Severe valve disease (e.g., critical aortic stenosis)
8. Cardiac conditions requiring an implanted cardiac device such as a pacemaker, defibrillator, or left ventricular assist device (for arrhythmia, congestive heart failure, etc.)
9. Untreated chest pain or angina
10. Patients with movement disorders (e.g., Parkinson's Disease)
11. History of Cerebral Vascular Accident (CVA), Transient Ischemic Attack (TIA), or seizures
12. Require home oxygen (O2) at rest or with exertion
13. End-stage renal disease (ESRD) requiring dialysis
14. Morbid obesity (BMI>35)
15. Patient undergoing cataract surgery in combination with any other ophthalmologic procedure
16. Patient requiring general anesthesia during cataract surgery due to the underlying characteristics of the existing cataract and/or anticipated complexity of the planned procedure

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction as assessed by the Iowa Satisfaction With Anesthesia Scale (ISAS) | 30 minutes, 1 day and 7 days after surgery
  The ISAS is a validated 11-question survey to find out how people feel about the sedation (i.e., monitored anesthesia care) they received during surgery that doesn't require general anesthesia. It asks about pain and overall feelings about the anesthesia care received. We will compare ISAS scores between patients who received oral sedation and patients who received placebo.

SECONDARY OUTCOMES:
Proportion of patients meeting eligibility criteria | Through study completion, an average of 1 year
  Number of patients meeting eligibility criteria divided by the total number of patients screened
Proportion of patients completing all study surveys after cataract surgery | Through study completion, an average of 1 year
  Number of patients completing all study surveys after cataract surgery divided by the number of patients enrolled in the study
Proportion of study patients who completed all required study procedures | Through study completion, an average of 1 year
  The number of study patients who completed all required study procedures (before and after surgery) divided by the number of patients enrolled in the study.
Incidence of sedation-related complications after surgery | 30 days after surgery
  The number of patients with a sedation-related complication divided by the number of patients enrolled in the study.
Quality of recovery after surgery using the Postoperative Quality of Recovery Scale (PQRS) | 30 minutes, 1 day and 7 days after surgery
  The PQRS is a 6-question survey that assesses the quality of recovery of patients after surgery. It evaluates multiple aspects of recovery, including physiological, pain, emotional, brain function, and activities of daily living domains.
Quality of recovery after surgery as measured by the Quality-of-Recovery-15 Questionnaire (QoR-15) | 1 day and 7 days after surgery
  The QoR-15 is a survey that has 15 questions and is used to see how patients feel after surgery and helps to understand the trajectory of recovery from surgery and anesthesia. The survey includes questions about mood, including if patients are feeling anxious or depressed.
Quality of recovery after surgery as measured by the Functional Recovery index (FRI) | 1 day and 7 days after surgery
  The FRI is a 14-question survey to check how well patients can do normal activities after surgery. It asks about things like pain, moving around, and daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine L Chen, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
This is a small single center pilot study so we do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Chen CL, Lin GA, Bardach NS, Clay TH, Boscardin WJ, Gelb AW, Maze M, Gropper MA, Dudley RA. Preoperative medical testing in Medicare patients undergoing cataract surgery. N Engl J Med. 2015 Apr 16;372(16):1530-8. doi: 10.1056/NEJMsa1410846. PMID 25875258
- [Background] Chen CL, Clay TH, McLeod S, Chang HP, Gelb AW, Dudley RA. A Revised Estimate of Costs Associated With Routine Preoperative Testing in Medicare Cataract Patients With a Procedure-Specific Indicator. JAMA Ophthalmol. 2018 Mar 1;136(3):231-238. doi: 10.1001/jamaophthalmol.2017.6372. PMID 29346472
- [Background] Liu YC, Wilkins M, Kim T, Malyugin B, Mehta JS. Cataracts. Lancet. 2017 Aug 5;390(10094):600-612. doi: 10.1016/S0140-6736(17)30544-5. Epub 2017 Feb 25. PMID 28242111
- [Background] Norregaard, J. C. Results from the International Cataract Surgery Outcomes Study. Acta Ophthalmologica Scandinavica 85, 5-32, doi:10.1111/j.1600-0420.2007.00937.x (2007).
- [Background] Kent, C. Cataract Surgery: Is an anesthesiologist necessary?, <https://www.reviewofophthalmology.com/article/cataract-surgery-is-an-anesthesiologist-necessary> (2009).
- [Background] Andrews, M. Anthem Calls On Eye Surgeons To Monitor Anesthesia During Cataract Surgery, <https://khn.org/news/anthem-calls-on-eye-surgeons-to-monitor-anesthesia-during-cataract-surgery/> (2018).
- [Background] Ianchulev T, Litoff D, Ellinger D, Stiverson K, Packer M. Office-Based Cataract Surgery: Population Health Outcomes Study of More than 21 000 Cases in the United States. Ophthalmology. 2016 Apr;123(4):723-8. doi: 10.1016/j.ophtha.2015.12.020. Epub 2016 Jan 22. PMID 26804760
- [Background] Zakrzewski PA, Friel T, Fox G, Braga-Mele R. Monitored anesthesia care provided by registered respiratory care practitioners during cataract surgery: a report of 1957 cases. Ophthalmology. 2005 Feb;112(2):272-7. doi: 10.1016/j.ophtha.2004.08.016. PMID 15691563
- [Background] Kent-Smith BT, Wallace GM. Routine cataract surgery without the presence of an anaesthetist. Clin Exp Ophthalmol. 2007 Aug;35(6):589. doi: 10.1111/j.1442-9071.2007.01553.x. No abstract available. PMID 17760646
- [Background] Murray P, Adams K, Haddad P, Murray N, O'Rourke M. The routine requirement for anaesthetists in local anaesthetic cataract surgery. Clin Exp Ophthalmol. 2007 Mar;35(2):195-6. doi: 10.1111/j.1442-9071.2006.01441.x. No abstract available. PMID 17362468
- [Background] Zakrzewski PA, Banashkevich AV, Friel T, Braga-Mele R. Monitored anesthesia care by registered respiratory therapists during cataract surgery: an update. Ophthalmology. 2010 May;117(5):897-902. doi: 10.1016/j.ophtha.2009.10.005. Epub 2010 Jan 15. PMID 20079927
- [Background] Basta B, Gioia L, Gemma M, Dedola E, Bianchi I, Fasce F, Beretta L. Systemic adverse events during 2005 phacoemulsifications under monitored anesthesia care: a prospective evaluation. Minerva Anestesiol. 2011 Sep;77(9):877-83. PMID 21878869
- [Background] Koolwijk J, Fick M, Selles C, Turgut G, Noordergraaf JI, Tukkers FS, Noordergraaf GJ. Outpatient cataract surgery: incident and procedural risk analysis do not support current clinical ophthalmology guidelines. Ophthalmology. 2015 Feb;122(2):281-7. doi: 10.1016/j.ophtha.2014.08.030. Epub 2014 Oct 22. PMID 25444350
- [Background] Katz J, Feldman MA, Bass EB, Lubomski LH, Tielsch JM, Petty BG, Fleisher LA, Schein OD. Injectable versus topical anesthesia for cataract surgery: patient perceptions of pain and side effects. The Study of Medical Testing for Cataract Surgery study team. Ophthalmology. 2000 Nov;107(11):2054-60. doi: 10.1016/s0161-6420(00)00359-6. PMID 11054331
- [Background] Katz J, Feldman MA, Bass EB, Lubomski LH, Tielsch JM, Petty BG, Fleisher LA, Schein OD; Study of Medical Testing for Cataract Surgery Study Team. Adverse intraoperative medical events and their association with anesthesia management strategies in cataract surgery. Ophthalmology. 2001 Oct;108(10):1721-6. doi: 10.1016/s0161-6420(01)00704-7. PMID 11581040
- [Background] Fukuoka H, Afshari NA. The impact of age-related cataract on measures of frailty in an aging global population. Curr Opin Ophthalmol. 2017 Jan;28(1):93-97. doi: 10.1097/ICU.0000000000000338. PMID 27820747
- [Background] American Society of Anesthesiologists. ASA Calls on Anthem to Rescind Its New Policy on Anesthesia for Cataract Surgery, <https://www.asahq.org/advocacy-and-asapac/fda-and-washington-alerts/washington-alerts/2018/02/asa-calls-on-anthem-to-rescind-its-new-policy-on-anesthesia-for-cataract-surgery?&ct=fd2b35b6cdb74e0b126f4539b73b56360091233e85002bc197d8049fa56b7a4253b022b37557ad25186cfc15475fa96cd09811e97c66fe62b04a1ec1298f82ef> (2018).
- [Background] American Academy of Ophthalmology. Pressure on Anthem Grows; Academy Keeps Pushing for Cataract-Surgery Anesthesia Coverage, 2018).
- [Background] Partridge JS, Harari D, Dhesi JK. Frailty in the older surgical patient: a review. Age Ageing. 2012 Mar;41(2):142-7. doi: 10.1093/ageing/afr182. PMID 22345294
- [Background] Hubbard RE, Story DA. Patient frailty: the elephant in the operating room. Anaesthesia. 2014 Jan;69 Suppl 1:26-34. doi: 10.1111/anae.12490. PMID 24303858
- [Background] McIsaac DI, MacDonald DB, Aucoin SD. Frailty for Perioperative Clinicians: A Narrative Review. Anesth Analg. 2020 Jun;130(6):1450-1460. doi: 10.1213/ANE.0000000000004602. PMID 32384334
- [Background] Kim DH, Patorno E, Pawar A, Lee H, Schneeweiss S, Glynn RJ. Measuring Frailty in Administrative Claims Data: Comparative Performance of Four Claims-Based Frailty Measures in the U.S. Medicare Data. J Gerontol A Biol Sci Med Sci. 2020 May 22;75(6):1120-1125. doi: 10.1093/gerona/glz224. PMID 31566201
- [Background] Kim DH, Schneeweiss S, Glynn RJ, Lipsitz LA, Rockwood K, Avorn J. Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index. J Gerontol A Biol Sci Med Sci. 2018 Jun 14;73(7):980-987. doi: 10.1093/gerona/glx229. PMID 29244057
- [Background] Hodge W, Horsley T, Albiani D, Baryla J, Belliveau M, Buhrmann R, O'Connor M, Blair J, Lowcock E. The consequences of waiting for cataract surgery: a systematic review. CMAJ. 2007 Apr 24;176(9):1285-90. doi: 10.1503/cmaj.060962. PMID 17452662
- [Background] Iroku-Malize T, Kirsch S. Eye Conditions in Older Adults: Cataracts. FP Essent. 2016 Jun;445:17-23. PMID 27348528
- [Background] Owsley C, McGwin G Jr, Sloane M, Wells J, Stalvey BT, Gauthreaux S. Impact of cataract surgery on motor vehicle crash involvement by older adults. JAMA. 2002 Aug 21;288(7):841-9. doi: 10.1001/jama.288.7.841. PMID 12186601
- [Background] Hillman, L. Phaco turns 50, <https://www.eyeworld.org/phaco-turns-50> (2017).
- [Background] Eke T, Thompson JR. Serious complications of local anaesthesia for cataract surgery: a 1 year national survey in the United Kingdom. Br J Ophthalmol. 2007 Apr;91(4):470-5. doi: 10.1136/bjo.2006.106005. Epub 2006 Nov 23. PMID 17124243
- [Background] Jefferis JM, Clarke MP, Taylor JP, Brittain KR. Challenges for the cataract surgeon treating people with dementia: a qualitative study exploring anesthetic choices. Clin Ophthalmol. 2014 Sep 26;8:1993-9. doi: 10.2147/OPTH.S69388. eCollection 2014. PMID 25328382
- [Background] Norregaard JC, Bernth-Petersen P, Bellan L, Alonso J, Black C, Dunn E, Andersen TF, Espallargues M, Anderson GF. Intraoperative clinical practice and risk of early complications after cataract extraction in the United States, Canada, Denmark, and Spain. Ophthalmology. 1999 Jan;106(1):42-8. doi: 10.1016/s0161-6420(99)90004-0. PMID 9917779
- [Background] Sharwood PL, Thomas D, Roberts TV. Adverse medical events associated with cataract surgery performed under topical anaesthesia. Clin Exp Ophthalmol. 2008 Dec;36(9):842-6. doi: 10.1111/j.1442-9071.2009.01924.x. PMID 19278479
- [Background] Stein JD, Grossman DS, Mundy KM, Sugar A, Sloan FA. Severe adverse events after cataract surgery among medicare beneficiaries. Ophthalmology. 2011 Sep;118(9):1716-23. doi: 10.1016/j.ophtha.2011.02.024. Epub 2011 Jun 2. PMID 21640382
- [Background] Rocha G, Turner C. Safety of cataract surgery under topical anesthesia with oral sedation without anesthetic monitoring. Can J Ophthalmol. 2007 Apr;42(2):288-94. PMID 17392854
- [Background] California Medical Association. CMA calls for investigation into Anthem restricting use of sedation during cataract surgery, <https://www.cmadocs.org/newsroom/news/view/ArticleID/21466/t/CMA-calls-for-investigation-into-Anthem-policy-restricting-use-of-sedation-during-cataract-surgery> (2018).
- [Background] Rosenfeld SI, Litinsky SM, Snyder DA, Plosker H, Astrove AW, Schiffman J. Effectiveness of monitored anesthesia care in cataract surgery. Ophthalmology. 1999 Jul;106(7):1256-60; discussion 1261. doi: 10.1016/S0161-6420(99)00705-8. PMID 10406602
- [Background] Dent E, Kowal P, Hoogendijk EO. Frailty measurement in research and clinical practice: A review. Eur J Intern Med. 2016 Jun;31:3-10. doi: 10.1016/j.ejim.2016.03.007. Epub 2016 Mar 31. PMID 27039014
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Whitlock EL, Whittington RA. The Frailty Syndrome: Anesthesiologists Must Understand More and Fear Less. Anesth Analg. 2020 Jun;130(6):1445-1448. doi: 10.1213/ANE.0000000000004789. No abstract available. PMID 32384332
- [Background] Fleisher LA, Fleischmann KE, Auerbach AD, Barnason SA, Beckman JA, Bozkurt B, Davila-Roman VG, Gerhard-Herman MD, Holly TA, Kane GC, Marine JE, Nelson MT, Spencer CC, Thompson A, Ting HH, Uretsky BF, Wijeysundera DN. 2014 ACC/AHA guideline on perioperative cardiovascular evaluation and management of patients undergoing noncardiac surgery: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines. Developed in collaboration with the American College of Surgeons, American Society of Anesthesiologists, American Society of Echocardiography, American Society of Nuclear Cardiology, Heart Rhythm Society, Society for Cardiovascular Angiography and Interventions, Society of Cardiovascular Anesthesiologists, and Society of Vascular Medicine Endorsed by the Society of Hospital Medicine. J Nucl Cardiol. 2015 Feb;22(1):162-215. doi: 10.1007/s12350-014-0025-z. No abstract available. PMID 25523415
- [Background] Aarons GA, Hurlburt M, Horwitz SM. Advancing a conceptual model of evidence-based practice implementation in public service sectors. Adm Policy Ment Health. 2011 Jan;38(1):4-23. doi: 10.1007/s10488-010-0327-7. PMID 21197565
- [Background] Glisson C, Landsverk J, Schoenwald S, Kelleher K, Hoagwood KE, Mayberg S, Green P; Research Network on Youth Mental Health. Assessing the organizational social context (OSC) of mental health services: implications for research and practice. Adm Policy Ment Health. 2008 Mar;35(1-2):98-113. doi: 10.1007/s10488-007-0148-5. Epub 2007 Dec 18. PMID 18085434
- [Background] Hays, D. G. & Singh, A. A. Qualitative inquiry in clinical and educational settings. (Guilford Press, 2012).
- [Background] Saunders B, Sim J, Kingstone T, Baker S, Waterfield J, Bartlam B, Burroughs H, Jinks C. Saturation in qualitative research: exploring its conceptualization and operationalization. Qual Quant. 2018;52(4):1893-1907. doi: 10.1007/s11135-017-0574-8. Epub 2017 Sep 14. PMID 29937585
- [Background] Francis JJ, Johnston M, Robertson C, Glidewell L, Entwistle V, Eccles MP, Grimshaw JM. What is an adequate sample size? Operationalising data saturation for theory-based interview studies. Psychol Health. 2010 Dec;25(10):1229-45. doi: 10.1080/08870440903194015. PMID 20204937
- [Background] Nilsen P. Making sense of implementation theories, models and frameworks. Implement Sci. 2015 Apr 21;10:53. doi: 10.1186/s13012-015-0242-0. PMID 25895742
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Guest, G., MacQueen, K. M. & Namey, E., E. Applied Thematic Analysis. (Sage Publications, 2011).
- [Background] MacQueen, K. M., McLellan, E., Kay, K. & Milstein, B. Codebook Development for Team-Based Qualitative Analysis. CAM Journal 10, 31-36, doi:10.1177/1525822x980100020301 (2016).
- [Background] Hays, D. G. & Singh, A. A. in Qualitative Inquiry in Clinical and Educational Settings Ch. 10, 292-336 (Guilford Press, 2011).
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459